CLINICAL TRIAL: NCT00281736
Title: A Phase II Study of HPPH Photodynamic Therapy for Treatment of High Grade Dysplasia, Carcinoma In-Situ or Early Intramucosal Adenocarcinoma in Barrett's Esophagus. Randomization to Two PDT Treatment Regimens of HPPH (2-1 [Hexyloxyethyl]-2devinylpyropheophorbide-a) and Light
Brief Title: Photodynamic Therapy in Treating Patients With Precancerous Esophageal Conditions or Early Stage Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441205; I 30404 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; stage 0 esophageal cancer; stage I esophageal cancer; precancerous condition
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Adenocarcinoma Of Esophagus | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive HPPH IV over 1 hour on day 1. Approximately 24 hours later, the lesion is exposed to laser light endoscopically.
  Interventions: Drug: HPPH
- Arm II (Experimental): Patients receive HPPH as in arm I, but at a higher dose, followed by laser light exposure.
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — Given IV

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as HPPH, that is absorbed by tumor cells. The drug becomes active when it is exposed to light, and kills tumor cells. HPPH may be effective in killing precancerous cells and tumor cells.

PURPOSE: This randomized phase II trial is studying how well photodynamic therapy with HPPH works in treating patients with precancerous esophageal conditions or stage 0 or stage I esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response in patients with high-grade dysplasia, carcinoma in situ, or early intramucosal adenocarcinoma of the esophagus and Barrett's esophagus treated with photodynamic therapy using HPPH.
* Determine the safety, in terms of toxicity to surrounding normal tissue, of this regimen in these patients.
* Determine the toxic effects of this regimen on surrounding normal tissue in these patients.
* Determine the incidence of adenocarcinoma in these patients after this treatment.
* Determine the magnitude and duration of increased skin sun sensitivity in patients treated with this regimen.
* Determine the minimal erythemal dose of this regimen in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to presence of intramucosal tumor (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive HPPH IV over 1 hour on day 1. Approximately 24 hours later, the lesion is exposed to laser light endoscopically.
* Arm II: Patients receive HPPH as in arm I, but at a higher dose, followed by laser light exposure.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 60 patients (30 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade dysplasia, carcinoma in situ, or early intramucosal adenocarcinoma of the esophagus

  * Stage 0 or N0, M0 primary or recurrent disease
* Diagnosis of Barrett's esophagus
* Ineligible for or refused surgical resection
* Requires endoscopy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 4,000/mm^3
* Platelet count ≥ 100,000/mm^3
* PT ≤ 1.5 times upper limit of normal (ULN)

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times ULN
* ALT ≤ 3 times ULN

Renal

* Creatinine ≤ 2 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No contraindication to endoscopy
* No other malignancy except nonmelanoma skin cancer or another cancer for which patient is deemed disease-free
* No porphyria or hypersensitivity to porphyrin or porphyrin-like compounds

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 1 month since prior chemotherapy
* No concurrent chemotherapy

Radiotherapy

* At least 1 month since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 1 month since prior Nd-YAG laser therapy
* At least 4 weeks since prior therapy for this disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 3 years

SECONDARY OUTCOMES:
Toxicity | 3 years
Response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hector R. Nava, MD, FACS, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States